CLINICAL TRIAL: NCT05504850
Title: The Feasibility and Acceptability of a Multicultural Healthy Diet (Anti-inflammatory Dietary Pattern) in Racial/Ethnic Minorities With Chronic Kidney Disease
Brief Title: Multicultural Healthy Diet in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-12753; K23DK124644-01A1 (NIH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants will receive the intervention (Other)
  Interventions: Other: Multicultural Health Diet

INTERVENTIONS:
Other: Multicultural Health Diet — The food-based components will be similar to the anti-inflammatory diet of the ongoing MHD study (NCT03240406), which emphasizes limiting animal and high saturated fat foods with focus on anti-inflammatory foods/food components specific to the cultural context of the participant. The diet will also be tailored to needs of the CKD population including a focus on lowering sodium intake. The intervention (dietary counseling) will be delivered by experienced kidney disease nutritionist.

SUMMARY:
This is a pilot intervention study to evaluate the feasibility and acceptability of a culturally-tailored anti-inflammatory diet intervention in participants with chronic kidney disease.

DETAILED DESCRIPTION:
This is a pilot pre-post comparison intervention study to evaluate the feasibility and acceptability of a culturally-tailored anti-inflammatory diet intervention. The study will recruit approximately 20 adult participants with chronic kidney disease (CKD) from nephrology clinics in the Bronx. The diet emphasizes limiting animal and high saturated fat foods with focus on anti-inflammatory foods/food components specific to the cultural context of the participant. The diet will also be tailored to needs of the CKD population including a focus on lowering sodium intake. The intervention will be delivered by an experienced nutritionist with expertise providing dietary counseling to patients with CKD. The investigative team will assess whether the diet is feasible, acceptable, and safe in patients with CKD through dietary intake assessments, questionnaires and serum biomarkers. Information from study will help inform the study design and intervention of a future large-scale, study aimed at improving CKD outcomes. The clinical site for the proposed study is at the Albert Einstein College of Medicine and Montefiore Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* CKD stage 3 (estimated glomerular filtration rate (eGFR) ≥ 30 ml/min/1.73m^2 to < 60 ml/min/1.73m^2)
* Residency in the Bronx
* Sufficient hearing, vision, and proficiency in English or Spanish to comprehend dietary counseling and low-level printed educational materials
* Provide written informed consent

Exclusion Criteria:

* History of hyperkalemia, or baseline serum potassium (K) > 4.8
* CKD stage 4 or higher estimated Glomerular Filtration Rate (eGFR) <30 ml/min/1.73 m^2
* Unwillingness/inability to make dietary changes or if primarily interested in weight loss as judged by discussion with the participant
* History of kidney transplant
* Poorly controlled diabetes (HbA1c >9%) or insulin use
* Any severe chronic illness, low literacy, or other serious condition that precludes making dietary changes and requires strict dietary restrictions or completion of study activities
* Plans to relocate out of New York City in the next 2 months
* Visual, auditory, or motor impairment that precludes completion of the assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of dietary intervention | From baseline to 2 months post baseline
  Feasibility of the dietary intervention will be assessed using the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool and the Energy-Adjusted Dietary Inflammatory Index Diet (E-DII®) platform. The ASA24® is a web-based tool that enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records, also known as food diaries. The EE-DII® is a scientific tool that quantifies the potential of a person's diet to cause inflammation, adjusting for total calorie intake for better accuracy. It assigns higher (positive) scores to pro-inflammatory diets (processed meats, sugary drinks) and lower (negative) scores to anti-inflammatory diets (leafy greens, fruits, fish). For this study scores at baseline (pre-intervention) will be compared to scores at 2 months using the E-DII®. The intervention will be considered feasible if ≥ 65% participants have a 2-point or more reduction from their baseline dietary inflammation score.
Acceptability of dietary intervention | 2 months post baseline
  Acceptability of the dietary intervention will be assessed using the Acceptability of the Multicultural Healthy Diet (MHD) in CKD questionnaire. Participants will be asked to rate acceptability based on five items regarding whether the dietary intervention met their approval; was appealing, whether they liked the diet, in general, and liked using herbs/spices that they had not used before; and would recommend the diet to family/friends. Responses to each item are rated on a 5-point ordinal scale: (Completely disagree, Disagree, Neither agree nor disagree, Agree or Completely agree). The number/percentage of participants selecting each category will be tabulated.

OTHER OUTCOMES:
Potassium level | 2 weeks after first session with nutritionist
  A serum potassium will be assessed 2 weeks after starting the diet as an added safety measure.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Johns, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Migliori M, Panichi V, de la Torre R, Fito M, Covas M, Bertelli A, Munoz-Aguayo D, Scatena A, Paoletti S, Ronco C. Anti-inflammatory effect of white wine in CKD patients and healthy volunteers. Blood Purif. 2015;39(1-3):218-223. doi: 10.1159/000371570. Epub 2015 Mar 31. PMID 25833063
- [Background] Nettleton JA, Steffen LM, Mayer-Davis EJ, Jenny NS, Jiang R, Herrington DM, Jacobs DR Jr. Dietary patterns are associated with biochemical markers of inflammation and endothelial activation in the Multi-Ethnic Study of Atherosclerosis (MESA). Am J Clin Nutr. 2006 Jun;83(6):1369-79. doi: 10.1093/ajcn/83.6.1369. PMID 16762949
- [Background] Mazidi M, Shivappa N, Wirth MD, Hebert JR, Kengne AP. Greater Dietary Inflammatory Index score is associated with higher likelihood of chronic kidney disease. Br J Nutr. 2018 Jul;120(2):204-209. doi: 10.1017/S0007114518001071. PMID 29947319
- [Background] Gupta J, Mitra N, Kanetsky PA, Devaney J, Wing MR, Reilly M, Shah VO, Balakrishnan VS, Guzman NJ, Girndt M, Periera BG, Feldman HI, Kusek JW, Joffe MM, Raj DS; CRIC Study Investigators. Association between albuminuria, kidney function, and inflammatory biomarker profile in CKD in CRIC. Clin J Am Soc Nephrol. 2012 Dec;7(12):1938-46. doi: 10.2215/CJN.03500412. Epub 2012 Sep 27. PMID 23024164
- [Background] Amdur RL, Feldman HI, Gupta J, Yang W, Kanetsky P, Shlipak M, Rahman M, Lash JP, Townsend RR, Ojo A, Roy-Chaudhury A, Go AS, Joffe M, He J, Balakrishnan VS, Kimmel PL, Kusek JW, Raj DS; CRIC Study Investigators. Inflammation and Progression of CKD: The CRIC Study. Clin J Am Soc Nephrol. 2016 Sep 7;11(9):1546-1556. doi: 10.2215/CJN.13121215. Epub 2016 Jun 23. PMID 27340285
- [Background] Shankar A, Sun L, Klein BE, Lee KE, Muntner P, Nieto FJ, Tsai MY, Cruickshanks KJ, Schubert CR, Brazy PC, Coresh J, Klein R. Markers of inflammation predict the long-term risk of developing chronic kidney disease: a population-based cohort study. Kidney Int. 2011 Dec;80(11):1231-8. doi: 10.1038/ki.2011.283. Epub 2011 Aug 24. PMID 21866089
- [Background] Miyamoto T, Carrero JJ, Stenvinkel P. Inflammation as a risk factor and target for therapy in chronic kidney disease. Curr Opin Nephrol Hypertens. 2011 Nov;20(6):662-8. doi: 10.1097/MNH.0b013e32834ad504. PMID 21825982
- [Background] Qian Q. Inflammation: A Key Contributor to the Genesis and Progression of Chronic Kidney Disease. Contrib Nephrol. 2017;191:72-83. doi: 10.1159/000479257. Epub 2017 Sep 14. PMID 28910792
- [Background] Ruiz S, Pergola PE, Zager RA, Vaziri ND. Targeting the transcription factor Nrf2 to ameliorate oxidative stress and inflammation in chronic kidney disease. Kidney Int. 2013 Jun;83(6):1029-41. doi: 10.1038/ki.2012.439. Epub 2013 Jan 16. PMID 23325084
- [Background] Vilaysane A, Chun J, Seamone ME, Wang W, Chin R, Hirota S, Li Y, Clark SA, Tschopp J, Trpkov K, Hemmelgarn BR, Beck PL, Muruve DA. The NLRP3 inflammasome promotes renal inflammation and contributes to CKD. J Am Soc Nephrol. 2010 Oct;21(10):1732-44. doi: 10.1681/ASN.2010020143. Epub 2010 Aug 5. PMID 20688930
- [Background] Christ A, Gunther P, Lauterbach MAR, Duewell P, Biswas D, Pelka K, Scholz CJ, Oosting M, Haendler K, Bassler K, Klee K, Schulte-Schrepping J, Ulas T, Moorlag SJCFM, Kumar V, Park MH, Joosten LAB, Groh LA, Riksen NP, Espevik T, Schlitzer A, Li Y, Fitzgerald ML, Netea MG, Schultze JL, Latz E. Western Diet Triggers NLRP3-Dependent Innate Immune Reprogramming. Cell. 2018 Jan 11;172(1-2):162-175.e14. doi: 10.1016/j.cell.2017.12.013. PMID 29328911
- [Background] Baer DJ, Judd JT, Clevidence BA, Tracy RP. Dietary fatty acids affect plasma markers of inflammation in healthy men fed controlled diets: a randomized crossover study. Am J Clin Nutr. 2004 Jun;79(6):969-73. doi: 10.1093/ajcn/79.6.969. PMID 15159225
- [Background] Lopez-Garcia E, Schulze MB, Meigs JB, Manson JE, Rifai N, Stampfer MJ, Willett WC, Hu FB. Consumption of trans fatty acids is related to plasma biomarkers of inflammation and endothelial dysfunction. J Nutr. 2005 Mar;135(3):562-6. doi: 10.1093/jn/135.3.562. PMID 15735094
- [Background] Lin J, Hu FB, Curhan GC. Associations of diet with albuminuria and kidney function decline. Clin J Am Soc Nephrol. 2010 May;5(5):836-43. doi: 10.2215/CJN.08001109. Epub 2010 Mar 18. PMID 20299364
- [Background] Odermatt A. The Western-style diet: a major risk factor for impaired kidney function and chronic kidney disease. Am J Physiol Renal Physiol. 2011 Nov;301(5):F919-31. doi: 10.1152/ajprenal.00068.2011. Epub 2011 Aug 31. PMID 21880837
- [Background] Lopez-Garcia E, Schulze MB, Fung TT, Meigs JB, Rifai N, Manson JE, Hu FB. Major dietary patterns are related to plasma concentrations of markers of inflammation and endothelial dysfunction. Am J Clin Nutr. 2004 Oct;80(4):1029-35. doi: 10.1093/ajcn/80.4.1029. PMID 15447916
- [Background] Farhadnejad H, Asghari G, Mirmiran P, Yuzbashian E, Azizi F. Micronutrient Intakes and Incidence of Chronic Kidney Disease in Adults: Tehran Lipid and Glucose Study. Nutrients. 2016 Apr 20;8(4):217. doi: 10.3390/nu8040217. PMID 27104561
- [Background] Huang X, Jimenez-Moleon JJ, Lindholm B, Cederholm T, Arnlov J, Riserus U, Sjogren P, Carrero JJ. Mediterranean diet, kidney function, and mortality in men with CKD. Clin J Am Soc Nephrol. 2013 Sep;8(9):1548-55. doi: 10.2215/CJN.01780213. Epub 2013 Jun 6. PMID 23744002
- [Background] Kim H, Caulfield LE, Garcia-Larsen V, Steffen LM, Grams ME, Coresh J, Rebholz CM. Plant-Based Diets and Incident CKD and Kidney Function. Clin J Am Soc Nephrol. 2019 May 7;14(5):682-691. doi: 10.2215/CJN.12391018. Epub 2019 Apr 25. PMID 31023928
- [Background] Ford ES, Giles WH, Myers GL, Rifai N, Ridker PM, Mannino DM. C-reactive protein concentration distribution among US children and young adults: findings from the National Health and Nutrition Examination Survey, 1999-2000. Clin Chem. 2003 Aug;49(8):1353-7. doi: 10.1373/49.8.1353. PMID 12881452
- [Background] Lakoski SG, Cushman M, Criqui M, Rundek T, Blumenthal RS, D'Agostino RB Jr, Herrington DM. Gender and C-reactive protein: data from the Multiethnic Study of Atherosclerosis (MESA) cohort. Am Heart J. 2006 Sep;152(3):593-8. doi: 10.1016/j.ahj.2006.02.015. PMID 16923436
- [Background] Inker LA, Schmid CH, Tighiouart H, Eckfeldt JH, Feldman HI, Greene T, Kusek JW, Manzi J, Van Lente F, Zhang YL, Coresh J, Levey AS; CKD-EPI Investigators. Estimating glomerular filtration rate from serum creatinine and cystatin C. N Engl J Med. 2012 Jul 5;367(1):20-9. doi: 10.1056/NEJMoa1114248. PMID 22762315
- [Background] Guasch-Ferre M, Hruby A, Salas-Salvado J, Martinez-Gonzalez MA, Sun Q, Willett WC, Hu FB. Olive oil consumption and risk of type 2 diabetes in US women. Am J Clin Nutr. 2015 Aug;102(2):479-86. doi: 10.3945/ajcn.115.112029. Epub 2015 Jul 8. PMID 26156740
- [Background] Bonaccio M, Bonanni AE, Di Castelnuovo A, De Lucia F, Donati MB, de Gaetano G, Iacoviello L; Moli-sani Project Investigators. Low income is associated with poor adherence to a Mediterranean diet and a higher prevalence of obesity: cross-sectional results from the Moli-sani study. BMJ Open. 2012 Nov 19;2(6):e001685. doi: 10.1136/bmjopen-2012-001685. Print 2012. PMID 23166131
- [Background] Bonaccio M, Di Castelnuovo A, Pounis G, Costanzo S, Persichillo M, Cerletti C, Donati MB, de Gaetano G, Iacoviello L; Moli-sani Study Investigators. High adherence to the Mediterranean diet is associated with cardiovascular protection in higher but not in lower socioeconomic groups: prospective findings from the Moli-sani study. Int J Epidemiol. 2017 Oct 1;46(5):1478-1487. doi: 10.1093/ije/dyx145. PMID 29040542
- [Background] Alisha Coleman-Jensen MPR, Christian A. Gregory, and Anita Singh. Household Food Security in the United States in 2017. US Department of Agriculture, Economic Research Service. 2018( ERR-256).
- [Background] Bower KM, Thorpe RJ Jr, Rohde C, Gaskin DJ. The intersection of neighborhood racial segregation, poverty, and urbanicity and its impact on food store availability in the United States. Prev Med. 2014 Jan;58:33-9. doi: 10.1016/j.ypmed.2013.10.010. Epub 2013 Oct 23. PMID 24161713
- [Background] Hager ER, Cockerham A, O'Reilly N, Harrington D, Harding J, Hurley KM, Black MM. Food swamps and food deserts in Baltimore City, MD, USA: associations with dietary behaviours among urban adolescent girls. Public Health Nutr. 2017 Oct;20(14):2598-2607. doi: 10.1017/S1368980016002123. Epub 2016 Sep 22. PMID 27652511
- [Background] Block JP, Scribner RA, DeSalvo KB. Fast food, race/ethnicity, and income: a geographic analysis. Am J Prev Med. 2004 Oct;27(3):211-7. doi: 10.1016/j.amepre.2004.06.007. PMID 15450633
- [Background] Sumlin LL, Brown SA. Culture and Food Practices of African American Women With Type 2 Diabetes. Diabetes Educ. 2017 Dec;43(6):565-575. doi: 10.1177/0145721717730646. Epub 2017 Sep 20. PMID 28929866
- [Background] van Rompay MI, McKeown NM, Castaneda-Sceppa C, Falcon LM, Ordovas JM, Tucker KL. Acculturation and sociocultural influences on dietary intake and health status among Puerto Rican adults in Massachusetts. J Acad Nutr Diet. 2012 Jan;112(1):64-74. doi: 10.1016/j.jada.2011.08.049. PMID 22389874
- [Background] Gibson AA, Sainsbury A. Strategies to Improve Adherence to Dietary Weight Loss Interventions in Research and Real-World Settings. Behav Sci (Basel). 2017 Jul 11;7(3):44. doi: 10.3390/bs7030044. PMID 28696389
- [Background] Beunza JJ, Toledo E, Hu FB, Bes-Rastrollo M, Serrano-Martinez M, Sanchez-Villegas A, Martinez JA, Martinez-Gonzalez MA. Adherence to the Mediterranean diet, long-term weight change, and incident overweight or obesity: the Seguimiento Universidad de Navarra (SUN) cohort. Am J Clin Nutr. 2010 Dec;92(6):1484-93. doi: 10.3945/ajcn.2010.29764. Epub 2010 Oct 20. PMID 20962161
- [Background] Howard BV, Manson JE, Stefanick ML, Beresford SA, Frank G, Jones B, Rodabough RJ, Snetselaar L, Thomson C, Tinker L, Vitolins M, Prentice R. Low-fat dietary pattern and weight change over 7 years: the Women's Health Initiative Dietary Modification Trial. JAMA. 2006 Jan 4;295(1):39-49. doi: 10.1001/jama.295.1.39. PMID 16391215
- [Background] Goraya N, Simoni J, Jo C, Wesson DE. Dietary acid reduction with fruits and vegetables or bicarbonate attenuates kidney injury in patients with a moderately reduced glomerular filtration rate due to hypertensive nephropathy. Kidney Int. 2012 Jan;81(1):86-93. doi: 10.1038/ki.2011.313. Epub 2011 Aug 31. PMID 21881553
- [Background] Goraya N, Simoni J, Jo CH, Wesson DE. Treatment of metabolic acidosis in patients with stage 3 chronic kidney disease with fruits and vegetables or oral bicarbonate reduces urine angiotensinogen and preserves glomerular filtration rate. Kidney Int. 2014 Nov;86(5):1031-8. doi: 10.1038/ki.2014.83. Epub 2014 Apr 2. PMID 24694986
- [Background] Johns TS, Brown DD, Litwin AH, Goldson G, Buttar RS, Kreimerman J, Lo Y, Reidy KJ, Bauman L, Kaskel F, Melamed ML. Group-Based Care in Adults and Adolescents With Hypertension and CKD: A Feasibility Study. Kidney Med. 2020 Apr 18;2(3):317-325. doi: 10.1016/j.xkme.2020.01.013. eCollection 2020 May-Jun. PMID 32734251

DOCUMENTS (1):
  • Informed Consent Form (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT05504850/ICF_000.pdf